CLINICAL TRIAL: NCT03629938
Title: Erişkinlerde Ayak Medial Longitudinal Ark Yüksekliğinin Değerlendirilmesi ve Sınıflandırılması
Brief Title: Evaluation and Classification of Foot Medial Longitudinal Arch Height in Adults
Status: Completed | Type: Observational
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 10840098-604.01.01-E.14217
Record Dates: First submitted 2018-07-21; First posted 2018-08-14 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2019-02

CONDITIONS: Pes Planus
Keywords: Feiss line; Medial longitudinal arch; Navicular drop; Pes planus
MeSH Terms: conditions — Flatfoot

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: evaluation — evaluation and classification of medial longitudinal arch height of foot in adults

SUMMARY:
The aim of the study is, to evaluate and classificate the medial longitudinal arch height in adult individuals. Aged between 18-40 years,350 adults who are voluntarily participate is going to be evaluate with Feiss Line(FL), Navicular Drop(ND) and Longitudinal Arch Angle(LAA) in subtalar neutral and resting position. Maximum, minimum values are going to be calculated. The 95% and 68% prediction intervals will be used as cut off limits.

DETAILED DESCRIPTION:
The aim of the study is, to evaluate and classificate the medial longitudinal arch height in adult individuals.

Aged between 18-40 years,350 adults who are voluntarily participate is going to be evaluate with Feiss Line(FL), Navicular Height(NH) and Longitudinal Arch Angle(LAA) in subtalar neutral and resting position. Maximum, minimum values are going to be calculated.

Participant's height, weight and foot length, from posterior aspect of calcaneus to the longest toe's tip, will be measured. Center of the medial malleolus, the navicular tuberosity and the head of the first metatarsal bone will be marked with a CD marker. With these landmarks in foot's relaxed position, neutrally, FL, NH and LAA will be measured by a ruler.

Feiss Line is a drawn line between the center of the medial malleolus to the head of the first metatarsal bone and then perpendicular line distance between this line and the navicular tuberosity will be drawn.The vertical line between the ground and the tubercle indicates Navicular Height. Center of goniometer placed at the navicular tuberosity then goniometer arms follow the medial malleolus and the head of the first metatarsal bone, degree between two arms indicates Longitudinal Arch Angle.

FL, NH, LAA mean values will be calculated. The 95% and 68% prediction intervals will be used as cut off limits.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-40
* Individuals who voluntarily agree to participate in the study

Exclusion Criteria:

* Those who have foot operation
* Foot trauma story which is causing an anatomic disorder

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Individuals that ages between 18-60 (adults), healthy male and female
Sampling Method: Probability Sample
Enrollment: 350 (Actual)
Dates: Start 2019-03-03 (Actual); Primary Completion 2019-04-14 (Actual); Study Completion 2019-05-28 (Actual)

PRIMARY OUTCOMES:
Medial longitudinal arch height | 10 days
  Navicular Height(NH) mean value, Center of the medial malleolus, the navicular tuberosity and the head of the first metatarsal bone will be marked with a CD marker. With these landmarks in foot's relaxed position, neutrally NH will be measured by a ruler.
  The vertical line between the ground and the tubercle indicates Navicular Height. After all data collection, the data will be entered into the Statistical Package for the Social Sciences (SPSS) and the average value calculated.

SECONDARY OUTCOMES:
Mean value differences between male and female | 10 days
  Mean value differences between male and female will be compared statistically with the Statistical Package for the Social Sciences (SPSS) program.
Correlation of arc measurements and standing length | 10 days
  Correlation of arc measurements and standing length will be correlated statistically with the Statistical Package for the Social Sciences (SPSS) program.
Medial Longitudinal Arch Cut Off Values | 10 days
  After average values calculated, cut off values will be generated from the data obtained from the arch height in standard, healthy individuals.

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa Sahin, PhD, Study Chair — Medipol University; Gizem Ergezen, MSc, Principal Investigator — Medipol University
Locations (1):
- Istanbul Medipol University, Istanbul, Beykoz, Turkey (Türkiye)